CLINICAL TRIAL: NCT03605381
Title: Morbidity Prevalence Estimate at Six Months Following a Stroke: A Cohort Study.
Brief Title: MORbidity PRevalence Estimate In StrokE
Acronym: MORe PREcISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aneurin Bevan University Health Board (Other)
Responsible Party: Principal Investigator, Dr Jonathan Hewitt, Clinical Senior Lecturer & Honorary Consultant Physician, Aneurin Bevan University Health Board
Other Study IDs: SP06; 03 ABUHB (Other Grant/Funding Number: Stroke Implementation Group (Wales))
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Stroke; CVA (Cerebrovascular Accident); CVA; Sequelae; Stroke, Ischemic; Stroke Hemorrhagic; Hemianopia; Hemiplegia; Hemiparesis; Aphasia; Cerebral Infarction; Intracerebral Hemorrhage; Anxiety; Depression; Dysphagia; Dysarthria; Hemispatial Neglect; Mild Cognitive Impairment
Keywords: Stroke; PROMs; Cohort
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Hemianopsia; Hemiplegia; Paresis; Aphasia; Cerebral Infarction; Cerebral Hemorrhage; Anxiety Disorders; Depression; Deglutition Disorders; Dysarthria; Perceptual Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Information regarding the likely progress of post-stroke symptoms is vitally important to stroke survivors to allow them to plan for the future and to adjust to life after stroke. Moreover, the prevalence of morbidity secondary to stroke is of central importance to Health Professionals to understand the prognosis of the disease in the patients under their care. Additionally, it will also allow commissioners of care, planners and third sector organisations to adapt to and answer the needs of a post-stroke population.

Currently, the data collected by national audit programmes are concentrated on what can be termed 'process or process of care' data. The utility of these data are in the ability to audit the care received by stroke survivors on stroke units against evidenced standards for care, thus ensuring evidence based practice. Nevertheless, process of care is only one form of measuring stroke unit care and the audit programmes collect some limited functional status data, data relating to risk-factor co-morbidities and treatment received data. Therefore, the scope of this study is to build on the minimum data set currently collected and to collect post-stroke data in domains not currently collected.

The International Consortium for Health Outcomes Measurement (ICHOM) takes important steps to collect data outside of process of care data such as a Patient Reported outcome data in their minimum outcome data set for stroke [currently under review].. Nevertheless, the ICHOM doesn't currently advocate the specific collection of data relating to cognitive impairment or emotional problems secondary to stroke. It is in these important aspects that this study will augment the data set currently advocated by ICHOM to collect data in the areas of cognitive impairment and emotional problems secondary to stroke.

Therefore, the aim of this study is to quantify the prevalence of morbidity at six months post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of stroke either;

  * Cerebral Infarct (ICD I63) [1]
  * Intracerebral Haemorrhage (ICD I61) [1]
  * Stroke, not specified as haemorrhage or infarction (ICD I64) [1]
* 18 years of age or older (≥ 18 years old)
* Received a clinically confirmed diagnosis of stroke within the previous 14 days (Stroke diagnosis ≤ 14 days)

Exclusion Criteria:

* Clinically confirmed diagnosis of any of the following

  * Transient Ischaemic Attack (ICD G45) [1]
  * Subarachnoid Haemorrhage (ICD I60) [1]
  * Any condition defined under ICD G93 e.g. Anoxic brain damage [1]
  * Patients receiving or eligible for Palliative Care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors admitted to stroke units across the UK
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Morbidity Secondary to Stroke | 6 months post-stroke
  The primary aim of this study is to quantify the prevalence of morbidity at six months post-stroke, measured using a PROM

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hewitt, MBBS, PhD, Principal Investigator — Cardiff University & Aneurin Bevan University Health Board
Locations (3):
- United Kingdom (3):
  - Ysbyty Ystrad Fawr, Ystrad Mynach, Caerphilly
  - Royal Gwent Hospital, Newport, Gwent
  - Prince Charles Hospital, Merthyr Tydfil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith A, Bains N, Copeland L, Pennington A, Carter B, Hewitt J. Morbidity Prevalence Estimate at 6 Months Following a Stroke: Protocol for a Cohort Study. JMIR Res Protoc. 2020 Jun 17;9(6):e15851. doi: 10.2196/15851. PMID 32512539